CLINICAL TRIAL: NCT06377384
Title: A Pilot and Feasibility Study Focusing on Lifestyle, Environmental Modifications, and Transdisciplinary Clinical Care for Children With Chronic Illness: Protocol for the FLIGHT Study
Brief Title: FLIGHT Study for Childhood Chronic Illness
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Documenting Hope Project (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DHP-33-FLIGHT
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Chronic Illnesses, Multiple
Keywords: children; chronic illness; total allostatic load; FLIGHT; functional medicine; environmental medicine; lifestyle medicine; root-cause medicine; personalized medicine
MeSH Terms: conditions — Multiple Chronic Conditions; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- FLIGHT Intervention (Experimental)
  Interventions: Other: FLIGHT Intervention

INTERVENTIONS:
Other: FLIGHT Intervention — Personalized and multimodality intervention focusing upon modifiable lifestyle factors, environmental modifications, and transdisciplinary clinical care.

SUMMARY:
The FLIGHT study is an open-label, single-arm, pilot and feasibility study of a personalized and multimodality intervention focusing upon modifiable lifestyle factors, environmental modifications, and transdisciplinary clinical care for children with chronic illness. A mixed methods outcomes evaluation will be performed. The primary goal of this study is to evaluate the most feasible and promising strategies to inform a more streamlined and scalable intervention in the future. Up to 14 participants may be enrolled, but fewer are expected to achieve the primary goal of the study.

ELIGIBILITY:
Inclusion Criteria:

* At least one guardian must have the ability to read and write English
* Participant and participant's caregiver must reside in the United States and live within the designated recruitment areas
* Verified completion of the CHIRP survey and consent to participate in the FLIGHT Study screening process
* Candidate's diagnosis(es) falls into one or more of the following categories:
* Immune/Autoimmune Conditions (for example: juvenile idiopathic arthritis, juvenile rheumatoid arthritis, asthma, eczema, atopic illness, allergies, Crohn's disease, ulcerative colitis, other gastrointestinal disorders, lupus, other autoimmune conditions)
* Conditions of Metabolic Dysregulation (for example: obesity/type 2 diabetes)
* Mood/Behavioral/Developmental Conditions (for example: autism spectrum disorders, ADHD/ADD, depression, obsessive-compulsive disorder, anxiety)
* Candidate is able to provide sufficient documentation of diagnoses, including validated/standardized diagnostic criteria in current use by specialists for each respective diagnosis, which have been performed by a professional with requisite experience or training

Exclusion Criteria:

* Candidate is a family member or close associate of any employees or board members of Epidemic Answers, members of the FLIGHT Study Team, or any advisors or clinicians associated with the FLIGHT Study
* Candidate is not able to provide documentation for proof of diagnoses
* Diagnosis with a condition that is severe enough to preclude participation in the intensive, multi-modal lifestyle intervention
* Caregiver(s) with health (e.g., serious chronic disease, disability, addiction) or other life circumstances (e.g., lack of transportation, shared custody of child) that preclude full participation in the intensive intervention
* External sources of environmental toxicants to the home or school environment that cannot be modified (e.g., high tension power line directly adjacent to home, coal-fired power plant within a ¼ mile of family's home)
* Inability to control/modify child's diet at daycare or with childcare provider
* Caregiver(s) anticipate a change of geographic location within two years
* Parent or caregiver has explicit belief that child's condition cannot be improved
* Caregiver(s) unwilling to make lifestyle changes, restrict candidate's non-essential technology use. prepare the majority of the family meals at home, replace personal and household products if indicated
* Caregiver(s) unwilling to have the candidate assessed by a team of doctors and/or healthcare practitioners including, but not limited to: physician, chiropractor, acupuncturist, optometrist, nutritionist, or other professionals recommend by the program
* Caregiver(s) unwilling to have the candidate participate in minimally invasive laboratory or non-laboratory assessments
* Caregiver(s) unwilling to have the candidate participate in required periodic video interviews, and other audio-visual documentation
* Candidate is pregnant
* Candidate has been convicted of a felony, is currently on probation, or in a juvenile detention center

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-06-07 (Actual)

PRIMARY OUTCOMES:
Total Load Index (TLI) | Baseline and 18 months
  The TLI is a measure of environmental, chemical, and social stressors that interact to contribute to chronic illness. There is no numeric score.

SECONDARY OUTCOMES:
Child Health Inventory for Resilience and Prevention (CHIRP) | Baseline, 3 months, 6 months, 9 months, 12 months, 15 months, 18 months
  Comprehensive survey evaluating total load of health stressors and supports influencing children. There is no numeric score.
Children's Sleep Habits Questionnaire (CSHQ) | Baseline, 3 months, 6 months, 9 months, 12 months, 15 months, 18 months
  Survey that assesses sleep. It consists of 35 items scored on a 1-3 point scale, with higher scores indicating worse sleep.
Vineland Adaptive Behavior Scale | Baseline, 9 months, 18 months
  Survey assessing developmental and other disorders. A standard score of 100 is considered average, with scores above 100 indicating strengths in adaptive behavior and scores below 100 indicating areas of difficulty.
Sensory Profile 2 | Baseline, 9 months, 18 months
  Survey assessing child's sensory processing patterns. There are 86 items. For each item, a score of 0 indicates that the individual's sensory processing is consistent with age-based norms. Positive scores suggest that the individual's sensory processing is better than age-based norms, while negative scores indicate that the individual's sensory processing is weaker than age-based norms.
Quick Environmental Exposure and Sensitivity Inventory (QEESI) | Baseline, 9 months, 18 months
  Survey that assesses environmental toxicants. The QEESI contains 50 items scored on a 0 to 10 scale with higher scores indicating greater environmental sensitivities.
Hayward Environmental Illness Severity Scale | Baseline, 9 months, 18 months
  Survey assessing impact of home environment on health. The survey consists of 22 questions with total score ranges from 0 to 100. Higher scores indicating greater severity of environmenal sensitivity symptoms.
Parenting Stress Index, 4th edition (PSI-4) | Baseline, 3 months, 6 months, 9 months, 12 months, 15 months, 18 months
  Survey assessing stress among parents. The PSI-4 contains 120 items with higher scores indicating greater levels of stress.
Beck Anxiety Inventory (BAI) | Baseline, 3 months, 6 months, 9 months, 12 months, 15 months, 18 months
  Survey assessing anxiety. The survey contains 21 items with scores ranging from 0 to 63. Higher scores indicate greater levels of anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Epidemic Answers, Windsor, Connecticut, United States